CLINICAL TRIAL: NCT06410768
Title: Evaluating the Feasibility of a Future Trial-based Economic Evaluation of a Multistage Shared Decision-making Program for the Treatment of Type 2 Diabetes Mellitus: a Pilot Study
Brief Title: Economic Evaluation of a Multistage Shared Decision-making Program for Type 2 Diabetes: a Pilot Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: METC2023-0114
Record Dates: First submitted 2024-04-22; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes mellitus; person-centered care; shared decision-making; pilot study; patient decision aid; economic evaluation
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): The intervention entails a multistage shared decision-making (SDM) program for type 2 diabetes mellitus (T2DM) that combines (1) an online PDA with (2) a preparatory consult for patients, and (3) interprofessional training in the PDA and SDM for healthcare professionals.
  Interventions: Behavioral: multistage shared decision-making program
- Control (No Intervention): Patients and healthcare professionals in the control practices will provide and receive usual care according to the national guidelines for T2DM of the Dutch College of General Practitioners (NHG). Participants in the control practices will not have access to the multistage SDM program.

INTERVENTIONS:
Behavioral: multistage shared decision-making program — The multistage shared decision-making program consists of 1) an online patient decision aid; 2) preparatory consult to provide patients with the knowledge and confidence to participate in shared decision-making; and 3) training to improve healthcare professionals' skills for shared decision-making.
  Arms: Intervention

SUMMARY:
Type 2 diabetes mellitus is a highly prevalent disease, affecting over a million Dutch citizens, leading to severe micro- and macrovascular complications, reduced quality of life, and high healthcare costs. Clinical guidelines recommend a person-centered approach to improve (health)outcomes. However, with rapidly increasing treatment options, both in terms of medication and lifestyle interventions, shared decision making (SDM) is challenging in practice. Therefore, researchers have developed a multistage SDM program consisting of an online patient decision aid for type 2 diabetes mellitus, training for healthcare professionals in SDM, and a preparatory consult to provide patients with the knowledge and confidence to participate in SDM. Strong evidence of (cost)-effectiveness is a key requirement to achieve broad implementation of this program. This pilot study represents an important initial step towards high-quality economic evaluation research, with a focus on the diversity of the study population, burden on participating healthcare practices, and feasibility of outcome measurement.

DETAILED DESCRIPTION:
Rationale: Previous randomized controlled trials researching the effects of shared decision-making (SDM) support through patient decision aids (PDAs) for type 2 diabetes mellitus (T2DM) experienced several challenges related to study procedures, resources, and study management. These challenges include difficulties in recruiting participants, understandability of questionnaires, timely recruitment, and inadvertent recruitment bias. Small-scale piloting is crucial to address uncertainties around the feasibility of trial methods and to refine the study procedures of a large-scale economic evaluation. This protocol outlines a pilot study aimed at evaluating the feasibility of a future trial-based economic evaluation of a multistage SDM program, including a PDA for T2DM in the Netherlands. By conducting a pilot study, the researchers aim to improve the quality of the intended trial-based economic evaluation.

Objectives: Researchers will conduct a pilot study focused on the following questions to prepare for an intended economic evaluation of our multistage SDM program for T2DM: 1) How to recruit and retain a representative sample of patients with T2DM in terms of sociodemographic and clinical background?; 2) How to support primary care practices in managing the challenges associated with study participation?; 3) How to feasibly measure relevant outcomes of SDM for T2DM using valid and reliable measurement instruments?

Study design: The multistage SDM program will be piloted in a cluster-randomized controlled trial using a mixed-methods approach. Four primary care practices will be included, of which two will be randomly assigned to the intervention group and two to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Is diagnosed with type 2 diabetes mellitus
* Eighteen years or older
* Need to decide on type 2 diabetes treatment based on the national guidelines
* Multiple treatment options (medication and/or lifestyle) are possible as judged by the healthcare professional
* Speak Dutch at a necessary level to complete questionnaires and ensure involvement in shared decision-making

Exclusion Criteria:

* Severe cognitive impairments that hamper shared decision-making

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Sample recruitment | 9 months
  Recruitment rates: how many patients were recruited on average for one month at one location.
  Time required to recruit to the target Sociodemographic and clinical characteristics
Sample retention | 9 months
  Retention rates: percentage of participants who completed the study
Consent rates | 9 months
  Consent rates: number of patients enrolled divided by number of eligible patients
Recruit to target | 9 months
  Time required to recruit to target sample size
Age (years) | Measured at baseline
  Age of participating patients in years. Patients are asked to complete a questionnaire at baseline that includes a question regarding their age.
Sex (self-reported questionnaire) | Measured at baseline
  Sex of participating patients. Patients are asked to complete a questionnaire at baseline that includes a question regarding their sex.
Country of birth (self-reported questionnaire) | Measured at baseline
  Country of birth of participating patients. Patients are asked to complete a questionnaire at baseline that includes a question regarding their country of birth.
Educational level (self-reported questionnaire) | Measured at baseline
  Educational level of participating patients. Patients are asked to complete a questionnaire at baseline that includes a question regarding their highest received diploma.
Financial (self-reported questionnaire) | Measured at baseline
  Make ends meet financially of participating patients. Patients are asked to complete a questionnaire at baseline that includes a question regarding their financial situation (i.e. whether they have (not) difficulties in making ends meet financially)
Work situation (self-reported questionnaire) | Measured at baseline
  Work situation of participating patients. Patients are asked to complete a questionnaire at baseline that includes a question regarding their work situation.
Duration of type 2 diabetes (self-reported questionnaire) | Measured at baseline
  Duration of diabetes of participating patients. Patients are asked to complete a questionnaire at baseline that includes a question regarding how many years they have type 2 diabetes.
Weight (kg) (self-reported questionnaire) | Measured at baseline
  Weight of participating patients in kg. Patients are asked to complete a questionnaire at baseline that includes a question regarding what their weight in kg is. This measure is used, in combination with height, to calculate their BMI.
Height (cm) (self-reported questionnaire) | Measured at baseline
  Height of participating patients in kg. Patients are asked to complete a questionnaire at baseline that includes a question regarding what their height in cm is. This measure is used, in combination with weight, to calculate their BMI.
Medication use (self-reported questionnaire) | Measured at baseline
  Medication use of participating patients in kg. Patients are asked to complete a questionnaire at baseline that includes a question regarding whether they use medication, and if so, whether they take oral medication or inject insulin.
Medication adherence measured with the Medication Adherence Report Scale (MARS) | Baseline, 3-months and 9-months follow-up
  Medication adherence measured with the Medication Adherence Report Scale (MARS) test. This test contains six statements regarding medication adherence and patients are asked to indicate whether the statements applies to them on a five point Likert Scale. Patients are asked to complete this test at baseline, 3 months and 9 months follow-up.
Health literacy (self-reported questionnaire) | Measured at baseline
  Health literacy of participating patients measured with the shortened version of the European Health Literacy Survey questionnaire (HLS-EU) Dutch questionnaire (6 questions)
Study management measured by conducting focus groups with participating healthcare professionals | Focus groups will be held at the end of patient inclusion period, 9-months
  Assessment of primary care practices' study management challenges (i.e. time constraints and capacity issues). This will be assessed by conducting focus groups with healthcare professionals from the participating general practices.
Patient decisional conflict measured with the decisional conflict scale (DCS) | Throughout implementation period, 9-months
  Decisional conflict measured with the 16-item decisional conflict scale (DCS). Patients will be asked to reflect on the treatment decision they made with their healthcare professional and respond to 16 statements in the DCS using a five-point Likert scale (ranging from completely agree to completely disagree). Besides a total score, the DCS includes five dimensions (i.e. information, support, clarification or values, certainty, and decision quality) with higher scores on a five-point scale indicating more decisional conflict. Patients are asked to complete this questionnaire at baseline, 3 months and 9 months follow-up.
Patient-rated level of shared decision-making measured with the 3-item CollaboRATE survey | Throughout implementation period, 9-months
  Patient-rated level of shared decision-making is measured by the 3-item CollaboRATE survey. The CollaboRATE survey assesses patients' perception of being informed and engaged in the decision-making steps on a scale of zero (no effort was made) to nine (every effort was made). Patients are asked to complete this questionnaire at baseline, 3 months and 9 months follow-up.
Patient-rated level of shared decision-making measured with the SDM-Q-9 questionnaire | Throughout implementation period, 9-months
  Patient-rated level of shared decision-making is measured by the SDM-Q-9 questionnaire. The SDM-Q-9 questionnaire measures the extent of shared decision-making durin a consultation between the patient and healthcare professional. This questionnaire consists of nine statements each describing a different step of the shared decision-making process. All items are scored on a six-point Likert scale from zero (completely disagree) to five (completely agree).
Healthcare professional level of shared decision-making measured with the SDM-Q-Doc questionnaire | Throughout implementation period, 9-months
  The SDM Q-Doc questionnaire (SDM-Q-9 adapted to the healthcare professional viewpoint) is used to measure the level of shared decision-making during a consultation from the perspective of a healthcare professional.
Patient knowledge measured with tailor-made questions | Measured at baseline
  Patient knowledge is measured with nine tailor-made multiple-choice questions assessing patients' understanding of the (risks and benefits of) glucose-lowering treatments.
Glycemic control obtained from general practitioner data | Baseline, 3-months and 9-months follow-up
  Glycemic control of participating patients will be obtained by obtaining HbA1c data from the general practitioner
Health-related quality of life measured with the EuroQol (EQ) 5 Dimension (5D) - 5 Level (5L) questionnaire | Baseline, 3-months and 9-months follow-up
  Health-related quality of life of participating patients will be measured with the Dutch EuroQol (EQ) 5 Dimension (5D) - 5 Level (5L) This measure facilitates utility calculations and includes the EQ-5D dimension and the EQ visual analog scale (EQ VAS). EQ-5D comprises five dimensions: mobility, self-care, pain, usual activities and anxiety. Each dimension is scored on a five-point Likert score (from no problems to extreme problems). The EQ VAS is used to assess the patient's self-reported health on a visual analog scale.
Medical consumption measured with the iMCQ | Baseline, 3-months and 9-months follow-up
  Medical consumption will be measured with an adapted version of the institute for Medical technology Assessment (iMTA) Medical Consumption Questionnaire (iMCQ).
Productivity costs measured with the iPCQ | Baseline, 3-months and 9-months follow-up
  Productivity costs will be measured with an adapted version of the institute for Medical technology Assessment (iMTA) Productivity Costs Questionnaire (iPCQ).
Understandability of measurement tools | Throughout the 9-month implementation period
  Sem-structured interviews with patients will be held to gain insight into the understandability of the measurement tools.

CONTACTS AND LOCATIONS:
Overall Officials: Arianne Elissen, PhD, Principal Investigator — Maastricht University
Locations (1):
- Care group Huisarts & Zorg, Gorinchem, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be made publicly available as a research article in a scientific journal. The protocol is under review.
Supporting Information: Study Protocol
Time Frame: The study protocol will be made publicly available as a research article in a scientific journal. The protocol is under review (April 2024).
Access Criteria: There will be no access criteria for the protocol (open access publication)

REFERENCES:
- [Background] Elwyn G, O'Connor A, Stacey D, Volk R, Edwards A, Coulter A, Thomson R, Barratt A, Barry M, Bernstein S, Butow P, Clarke A, Entwistle V, Feldman-Stewart D, Holmes-Rovner M, Llewellyn-Thomas H, Moumjid N, Mulley A, Ruland C, Sepucha K, Sykes A, Whelan T; International Patient Decision Aids Standards (IPDAS) Collaboration. Developing a quality criteria framework for patient decision aids: online international Delphi consensus process. BMJ. 2006 Aug 26;333(7565):417. doi: 10.1136/bmj.38926.629329.AE. Epub 2006 Aug 14. PMID 16908462
- [Background] ElSayed NA, Aleppo G, Aroda VR, Bannuru RR, Brown FM, Bruemmer D, Collins BS, Hilliard ME, Isaacs D, Johnson EL, Kahan S, Khunti K, Leon J, Lyons SK, Perry ML, Prahalad P, Pratley RE, Seley JJ, Stanton RC, Gabbay RA, on behalf of the American Diabetes Association. 9. Pharmacologic Approaches to Glycemic Treatment: Standards of Care in Diabetes-2023. Diabetes Care. 2023 Jan 1;46(Suppl 1):S140-S157. doi: 10.2337/dc23-S009. PMID 36507650
- [Background] Davies MJ, Aroda VR, Collins BS, Gabbay RA, Green J, Maruthur NM, Rosas SE, Del Prato S, Mathieu C, Mingrone G, Rossing P, Tankova T, Tsapas A, Buse JB. Management of hyperglycaemia in type 2 diabetes, 2022. A consensus report by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetologia. 2022 Dec;65(12):1925-1966. doi: 10.1007/s00125-022-05787-2. Epub 2022 Sep 24. PMID 36151309
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America. Crossing the Quality Chasm: A New Health System for the 21st Century. Washington (DC): National Academies Press (US); 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK222274/ PMID 25057539
- [Background] Stacey D, Legare F, Col NF, Bennett CL, Barry MJ, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L, Wu JH. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2014 Jan 28;(1):CD001431. doi: 10.1002/14651858.CD001431.pub4. PMID 24470076
- [Background] Stacey D, Suwalska V, Boland L, Lewis KB, Presseau J, Thomson R. Are Patient Decision Aids Used in Clinical Practice after Rigorous Evaluation? A Survey of Trial Authors. Med Decis Making. 2019 Oct;39(7):805-815. doi: 10.1177/0272989X19868193. Epub 2019 Aug 17. PMID 31423911
- [Background] Kellar I, Mann E, Kinmonth AL, Prevost AT, Sutton S, Marteau TM. Can informed choice invitations lead to inequities in intentions to make lifestyle changes among participants in a primary care diabetes screening programme? Evidence from a randomized trial. Public Health. 2011 Sep;125(9):645-52. doi: 10.1016/j.puhe.2011.05.010. Epub 2011 Jul 20. PMID 21764087
- [Background] Branda ME, LeBlanc A, Shah ND, Tiedje K, Ruud K, Van Houten H, Pencille L, Kurland M, Yawn B, Montori VM. Shared decision making for patients with type 2 diabetes: a randomized trial in primary care. BMC Health Serv Res. 2013 Aug 8;13:301. doi: 10.1186/1472-6963-13-301. PMID 23927490
- [Background] Mathers N, Ng CJ, Campbell MJ, Colwell B, Brown I, Bradley A. Clinical effectiveness of a patient decision aid to improve decision quality and glycaemic control in people with diabetes making treatment choices: a cluster randomised controlled trial (PANDAs) in general practice. BMJ Open. 2012 Nov 5;2(6):e001469. doi: 10.1136/bmjopen-2012-001469. Print 2012. PMID 23129571
- [Background] Mullan RJ, Montori VM, Shah ND, Christianson TJ, Bryant SC, Guyatt GH, Perestelo-Perez LI, Stroebel RJ, Yawn BP, Yapuncich V, Breslin MA, Pencille L, Smith SA. The diabetes mellitus medication choice decision aid: a randomized trial. Arch Intern Med. 2009 Sep 28;169(17):1560-8. doi: 10.1001/archinternmed.2009.293. PMID 19786674
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] van Teijlingen E, Hundley V. The importance of pilot studies. Nurs Stand. 2002 Jun 19-25;16(40):33-6. doi: 10.7748/ns2002.06.16.40.33.c3214. PMID 12216297
- [Background] Black SA. Diabetes, diversity, and disparity: what do we do with the evidence? Am J Public Health. 2002 Apr;92(4):543-8. doi: 10.2105/ajph.92.4.543. PMID 11919048
- [Background] Brodaty H, Gibson LH, Waine ML, Shell AM, Lilian R, Pond CD. Research in general practice: a survey of incentives and disincentives for research participation. Ment Health Fam Med. 2013 Sep;10(3):163-73. PMID 24427184
- [Background] McKinley N, McCain RS, Convie L, Clarke M, Dempster M, Campbell WJ, Kirk SJ. Resilience, burnout and coping mechanisms in UK doctors: a cross-sectional study. BMJ Open. 2020 Jan 27;10(1):e031765. doi: 10.1136/bmjopen-2019-031765. PMID 31988223
- [Background] West CP, Dyrbye LN, Shanafelt TD. Physician burnout: contributors, consequences and solutions. J Intern Med. 2018 Jun;283(6):516-529. doi: 10.1111/joim.12752. Epub 2018 Mar 24. PMID 29505159
- [Background] Tichler A, Hertroijs DFL, Ruwaard D, Brouwers MCGJ, Hiligsmann M, de Jong JD, Elissen AMJ. Preferred Conversation Topics with Respect to Treatment Decisions Among Individuals with Type 2 Diabetes. Patient Prefer Adherence. 2023 Mar 17;17:719-729. doi: 10.2147/PPA.S397647. eCollection 2023. PMID 36960182
- [Background] Legare F, Ratte S, Gravel K, Graham ID. Barriers and facilitators to implementing shared decision-making in clinical practice: update of a systematic review of health professionals' perceptions. Patient Educ Couns. 2008 Dec;73(3):526-35. doi: 10.1016/j.pec.2008.07.018. Epub 2008 Aug 26. PMID 18752915
- [Derived] Tichler A, Hertroijs DFL, van Mastrigt GAPG, Brouwers MCGJ, Ruwaard D, Elissen AMJ. Evaluating the feasibility of study methods for a future trial-based economic evaluation of a multistage shared decision-making program for type 2 diabetes mellitus: Protocol for a cluster-randomized controlled pilot study. PLoS One. 2025 Aug 5;20(8):e0300944. doi: 10.1371/journal.pone.0300944. eCollection 2025. PMID 40763135